CLINICAL TRIAL: NCT06250283
Title: Resveratrol for the Prevention of Bone Loss in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2043372; U54GM104941 (NIH)
Record Dates: First submitted 2024-01-18; First posted 2024-02-09 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-10

CONDITIONS: Low Bone Mass
Keywords: Resveratrol; Bone Health; Women Health
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): Dietary Supplement: Resveratrol (500 mg) + 500 mg calcium and 400 IU vitamin D3
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Dietary Supplement: Placebo (500 mg) + 500 mg calcium and 400 IU vitamin D3
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol (500 mg)
  Arms: Resveratrol
Dietary Supplement: Placebo — Placebo (500 mg)
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether daily supplementation of resveratrol would improve bone health in postmenopausal women.

DETAILED DESCRIPTION:
We plan to enroll and screen 68 women, with an estimated 34 qualifying women will be randomly assigned to two groups: 1) the placebo group and 2) the resveratrol group. The resveratrol group will receive 500 mg resveratrol daily for 24 weeks, and placebo group will receive placebo pills. Both groups will receive 500 mg calcium plus 400 IU vitamin D daily.

Blood and urinary biomarkers of bone metabolism will be assessed at baseline and after 12 and 24 weeks intervention. Bone mineral density will be assessed using dual-energy X-ray absorptiometry at baseline and after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1 to 10 years postmenopausal women with low bone mass

Exclusion Criteria:

* Osteoporosis
* Taking blood thinners, endocrine, or neuroactive drugs
* Hormone therapy
* Diagnosed: Metabolic bone disease, renal disease, kidney stones, cancer, cardiovascular disease, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease
* Severe menopausal symptoms, serious mood alterations, sleep disturbances
* Abnormal uterine bleeding, endometriosis, pelvic inflammatory disease
* Endometrial polyps, and significant uterine fibroids
* Smokers (≥ 20 cigarettes per day)
* BMI <20 and > 30 kg/m2
* Intolerance or allergic reaction to resveratrol, microcrystalline cellulose, grapes, red wine, or blueberries

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Bone biomarker | Bone marker will be assessed before and after 12 weeks and 24 weeks intervention
  25-hydroxy vitamin D3
Bone biomarker | Bone marker will be assessed before and after 12 weeks and 24 weeks intervention
  Alkaline phosphatase
Bone biomarker | Bone marker will be assessed before and after 12 weeks and 24 weeks intervention
  Osteocalcin
Bone biomarker | Bone marker will be assessed before and after 12 weeks and 24 weeks intervention
  Deoxypyridinoline
Bone biomarker | Bone marker will be assessed before and after 12 weeks and 24 weeks intervention
  C-terminal telopeptide type I collagen

SECONDARY OUTCOMES:
Bone mineral density | Bone mineral density will be assessed before and after 24 weeks intervention
  Lumbar spine, hip, forearm, and whole-body bone mineral density and bone mineral content

CONTACTS AND LOCATIONS:
Overall Officials: Sheau Ching Chai, PhD, RD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No